CLINICAL TRIAL: NCT03916822
Title: Validating Cell-based Assays for ABMR After Renal Transplantation
Brief Title: Cell-based Assays for Antibody-mediated Transplant Rejection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Plexision (Industry)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 00033434
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Antibody-Mediated Graft Rejection
Keywords: Antibody mediated Rejection; Renal Transplantation; Adults; CD154; B-cells; B-cell subsets; alloantigen-specific

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood leukocytes extracted from whole blood samples will be retained in liquid nitrogen for repeat testing or quality assessment until study results are public
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ABMR: Biopsy-proven ABMR-Banff criteria, with or without Complement binding donor-specific anti-HLA antibodies
  Interventions: Diagnostic Test: Alloantigen-specific B-cells
- TCMR: Biopsy-proven TCMR-Banff 1A, 1B, 2 and 3
  Interventions: Diagnostic Test: Alloantigen-specific B-cells
- No Rejection: Biopsy-proven, or clinical criteria
  Interventions: Diagnostic Test: Alloantigen-specific B-cells

INTERVENTIONS:
Diagnostic Test: Alloantigen-specific B-cells — Alloantigen-specific B-cells which express CD154 and their subsets which also co-express cytokines, memory and naive markers, and additional derivatives of these markers will be measured with flow cytometry

SUMMARY:
Goal: The goal of this study is to validate blood tests, which can detect antibody-mediated rejection (ABMR) after renal transplantation. These cell based assays measure CD154-expressing alloantigen-specific B-cells and their subsets in peripheral blood of adult renal transplant recipients. Thirty recipients will be enrolled at two transplant centers, 10 each with ABMR, T-cell mediated rejection (TCMR), and no rejection. Each subject will be sample twice, before and after rejection. Donor-specific anti-HLA antibodies will also be measured with single antigen beads.

DETAILED DESCRIPTION:
This cross-sectional open label study will evaluate whether alloantigen-specific B-cells and their subsets which express CD154 are associated with antibody-mediated rejection after first time renal transplantation in adult recipients.

Control groups include adult renal transplant recipients with T-cell-mediated rejection, and without rejection of any type.

Alloantigen-specific B-cells will be measured after stimulation of recipient peripheral blood leukocytes with those from corresponding donor and HLA-non-identical reference cells.

Thirty total subjects will be enrolled after IRB-approved informed consent, 15 at each of two sites. These subjects will include ten each with biopsy-proven ABMR and TCMR and ten with no rejection.

Each subject will be sampled twice, before and after treatment rejection, at intervals no less than 30 days, and not to exceed 90 days.

B-cells subsets will include those that also express cytokines, and those that are categorized as memory or naive, and their isotope switched or unswitched subsets, transitional B-cells or plasmablasts, etc.

ELIGIBILITY:
Inclusion Criteria:

* IRB-approved informed consent.
* Adults (>18 yr to 70 years)
* Primary renal transplant recipients with biopsy-proven ABMR, TCMR or recipients with no rejection

Exclusion Criteria:

* Lack of informed consent
* Concomitant BK virus infection
* Vulnerable populations including children <18 yr, pregnant women, and prisoners

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults who have received primary renal transplants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-06-14 (Estimated); Study Completion 2021-08-14 (Estimated)

PRIMARY OUTCOMES:
Antibody-mediated rejection | up to 90 days per subject
  Biopsy-proven antibody-mediated rejection after primary renal transplantation

SECONDARY OUTCOMES:
T-cell mediated rejection (TCMR) | up to 90 days per subject
  Biopsy-proven TCMR after primary renal transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Sindhi, MD, Study Director — Plexision
Locations (2):
- United States (2):
  - Erie County Medical Center, Buffalo, New York
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No
IPD will be retained at enrollment sites, Results of testing samples, and related de-identified data of the subject will be summarized and shared with all investigators of this study, and reported in publications